CLINICAL TRIAL: NCT05506540
Title: A Phase 1, First-in-human, 2-part, Randomized, Double-blind, Placebo-controlled, Parallel-group, Single Ascending Dose and Multiple Ascending Dose (SAD/MAD) Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ENN0403 in Healthy Adult Subjects
Brief Title: A First-in-human Single Ascending Dose/Multiple Ascending Dose Study of ENN0403 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EnnovaBio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ENN0403-P1-01
Record Dates: First submitted 2022-08-09; First posted 2022-08-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (10):
- Single Ascending Dose, ENN0403 1 mg (Experimental): Single oral use of ENN0403 at dose level 1 mg, in fasted state.
  Interventions: Drug: ENN0403 1mg
- Single Ascending Dose, ENN0403 4 mg (Experimental): Single oral use of ENN0403 at dose level 4 mg, in fasted state.
  Interventions: Drug: ENN0403 4mg
- Single Ascending Dose, ENN0403 10 mg (Experimental): Single oral use of ENN0403 at dose level 10 mg, in fasted state.
  Interventions: Drug: ENN0403 10mg
- Single Ascending Dose, ENN0403 20 mg (Experimental): Single oral use of ENN0403 at dose level 20 mg, in fasted state.
  Interventions: Drug: ENN0403 20mg
- Single Ascending Dose, ENN0403 30 mg (Experimental): Single oral use of ENN0403 at dose level 30 mg, in fasted state.
  Interventions: Drug: ENN0403 30mg
- Single Ascending Dose, ENN0403 20 mg (Fed) (Experimental): Single oral use of ENN0403 at dose level 30 mg, after high calorie and high-fat breakfast meal.
  Interventions: Drug: ENN0403 20mg (Fed)
- Multiple Ascending Dose, ENN0403 6 mg (Experimental): ENN0403 capsules for oral administration, 6 mg QD X 14 Days
  Interventions: Drug: ENN0403 6mg QD X 14 Days
- Multiple Ascending Dose, ENN0403 12 mg (Experimental): ENN0403 capsules for oral administration, 12 mg QD X 14 Days
  Interventions: Drug: ENN0403 12mg QD X 14 Days
- Multiple Ascending Dose, ENN0403 20 mg (Experimental): ENN0403 capsules for oral administration, 20 mg QD X 14 Days
  Interventions: Drug: ENN0403 20mg QD X 14 Days
- Single/Multiple Ascending Dose, placebo capsules for oral adminstration (Placebo Comparator): Placebo capsules for oral administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ENN0403 1mg — ENN0403 capsules for oral use
  Arms: Single Ascending Dose, ENN0403 1 mg
Drug: ENN0403 4mg — ENN0403 capsules for oral use
  Arms: Single Ascending Dose, ENN0403 4 mg
Drug: ENN0403 10mg — ENN0403 capsules for oral use
  Arms: Single Ascending Dose, ENN0403 10 mg
Drug: ENN0403 20mg — ENN0403 capsules for oral use
  Arms: Single Ascending Dose, ENN0403 20 mg
Drug: ENN0403 30mg — ENN0403 capsules for oral use
  Arms: Single Ascending Dose, ENN0403 30 mg
Drug: ENN0403 20mg (Fed) — ENN0403 capsules for oral use
  Arms: Single Ascending Dose, ENN0403 20 mg (Fed)
Drug: ENN0403 6mg QD X 14 Days — ENN0403 capsules for oral use
  Arms: Multiple Ascending Dose, ENN0403 6 mg
Drug: ENN0403 12mg QD X 14 Days — ENN0403 capsules for oral use
  Arms: Multiple Ascending Dose, ENN0403 12 mg
Drug: ENN0403 20mg QD X 14 Days — ENN0403 capsules for oral use
  Arms: Multiple Ascending Dose, ENN0403 20 mg
Drug: Placebo — Placebo capsules for oral use
  Arms: Single/Multiple Ascending Dose, placebo capsules for oral adminstration

SUMMARY:
This is a FIH, randomized, double- blind, placebo-controlled, dose -escalation study to investigate the safety, tolerability, PK, and PD of ENN0403 after single and multiple oral dose administration in healthy adult subjects. The study will include 2 parts which will proceed in a parallel staggered manner: Part A, a single ascending dose (SAD) study and Part B, a multiple ascending dose (MAD) study.

Approximately 80 healthy adult subjects will be enrolled at a single site in Australia, in up to 6 cohorts in Part A (SAD study), including a Food Effect (FE) study, and up to 4 cohorts in Part B (MAD study). Part A is for the single dose use of IP, while Part B is once daily use for 14 consecutive days. Each cohort will include 8 subjects (6 receiving ENN0403 and 2 receiving placebo). Each subject will be enrolled in only 1 cohort and receive only one dose regimen in this study.

Dosing will be escalated in a sequential fashion, contingent on a review of safety, tolerability, and available PK data of the previous dose level by a Safety Review Committee (SRC). The proposed dose levels/ dosing frequency of ENN0403 may be adjusted over the course of the whole study and cohorts may be added or removed depending on the emerging safety, tolerability, and available PK data.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent.
* 18 to 55 years old (inclusive).
* BMI of 18 to 30 kg/m2 (inclusive); body weight >50 to <100 kg for male subjects or >45 to <100 kg for female subjects.
* Computerized (12-lead) ECG recording without signs of clinically relevant pathology or showing no clinically relevant deviations as judged by the PI.
* Test negative for COVID-19.
* Test negative for HBsAg, anti-HBc, anti-hepatitis C virus (HCV) antibodies, anti-human immuno deficiencyvirus (HIV) 1 and 2 antibodies, and tuberculosis.
* Have a negative urine drug screen and a negative alcohol breath test.
* Nonsmoker or occasional smoker and willingness to refrain from smoking during study.
* Ability and willingness to abstain from alcohol during study.
* not pregnant, not breastfeeding; apply contraception methods for child-bearing potential subjects.

Exclusion Criteria:

* History of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal,cardiovascular, hepatic, psychiatric, neurologic, or allergic disease in the opinion of the Investigator within 12 months prior to Screening.
* Any disease or take any medication that affects IP absorption, distribution, metabolism, and excretion.3. Family history of sudden death or of congenital prolongation of the QTc interval or known congenital prolongation of the QTc interval or any clinical condition known to prolong the QTc interval.
* Presence of malignancy including hematological malignancies. Subjects with a history of basal cell or squamous cell carcinoma that has been treated with no evidence of recurrence within 3 years of Screening will be allowed for inclusion, as judged by the Investigator.
* Any current active infections, including localized infections, or any recent history (within 1 week prior to IP administration) of active infections, cough or fever; or a history of recurrent or chronic infections.
* In the 12-lead ECG assessment, QTcF >450 ms for male subjects or >470 ms for female subjects.7. Estimated glomerular fltration rate <90 mL /min (using the Cockcroft-Gault formula) at Screening.
* ALT or aspartate aminotransferase>1.5ULN.
* Have received any live vaccines (bacterial or viral) within 12 weeks prior to Screening or intend to receive a live vaccine during the study period or within 30 days after the last dose of the IP.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment emergent adverse events (TEAE) following ENN0403 administration | From first dose of ENN0403 administration till 7 days after last dose of ENN0403 administration.

SECONDARY OUTCOMES:
Maximum Plasma Concentration [Cmax] | Single Ascending Dose (SAD) part: up to Day 4, 72 hours post dose; Multiple Ascending Dose (MAD) part: up to Day 17, 72 hours post last dose
  Cmax is the maximum measured concentration of ENN0403 in plasma after oral administration
Area Under the Curve [AUC] | Single Ascending Dose (SAD) part: up to Day 4, 72 hours post dose; Multiple Ascending Dose (MAD) part: up to Day 17, 72 hours post last dose
  AUC is the area under the concentration-time curve of ENN0403 in plasma after oral administration

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX Clinical Research Pty Ltd, Adelaide, Adelaide, Australia

IPD SHARING:
Plan to Share IPD: No